CLINICAL TRIAL: NCT01736176
Title: An Open-Label, Two Part, Multicenter Study to Assess the Safety and Efficacy of Levodopa-Carbidopa Intestinal Gel (LCIG) for the Treatment of Non-Motor Symptoms in Subjects With Advanced Parkinson's Disease
Brief Title: A Study to Assess the Safety and Efficacy of Levodopa-carbidopa Intestinal Gel (LCIG) for the Treatment of Non-motor Symptoms in Patients With Advanced Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M12-920
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Advanced Parkinson's Disease
Keywords: Safety and efficacy; Advanced Parkinson's disease; levodopa-carbidopa intestinal gel,; carbidopa; levodopa; Non-Motor Symptom Scale
MeSH Terms: interventions — carbidopa, levodopa drug combination; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levodopa-Carbidopa Intestinal Gel (Experimental): Participants had the PEG-J tube placement procedure performed on Study Day 1 and, at the discretion of the investigator, began initiation and titration of LCIG infusion. Dosing was determined individually. The starting total daily dose of LCIG was based solely on the daily dose of the oral levodopa taken immediately prior to Study Day 1 and was adjusted to obtain the optimal clinical response for the individual participant.
  Participants received treatment for up to 60 weeks; participants who completed their Week 60 visit before LCIG was commercially available had the option to extend their LCIG therapy, if in the opinion of the investigator, the participant would benefit from continued LCIG treatment.
  Interventions: Drug: Levodopa-Carbidopa Intestinal Gel; Procedure: Percutaneous Endoscopic Gastrostomy with Jejunal Extension (PEG-J); Drug: Levodopa-carbidopa Immediate Release (LC-IR) Tablets

INTERVENTIONS:
Drug: Levodopa-Carbidopa Intestinal Gel — Levodopa-carbidopa intestinal gel (LCIG) for upper-intestinal infusion is a suspension of levodopa (20 mg/mL) and carbidopa monohydrate (5 mg/mL) in an aqueous gel, administered continuously by a portable pump via a percutaneous endoscopic gastrojejunostomy (PEG-J) tube.
  The rate of LCIG infusion was expected to be within the range of 1 to 10 mL/hour (20 to 200 mg of levodopa/hour) in most instances over a period of 16 consecutive hours.
  Other Names: Duopa; Carbidopa-levodopa enteral suspension (CLES)
Procedure: Percutaneous Endoscopic Gastrostomy with Jejunal Extension (PEG-J)
Drug: Levodopa-carbidopa Immediate Release (LC-IR) Tablets — After LCIG initiation, participants could take prescribed oral levodopa-carbidopa immediate or continuous release (i.e., oral LC prescribed by the investigator) for nighttime use.

SUMMARY:
The primary objective of this study is to evaluate change in non-motor symptoms from baseline to Week 12 as measured by the Non-Motor Symptom Scale total score.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a diagnosis of idiopathic Parkinson's disease (PD) according to the United Kingdom Parkinson's Disease Society (UKPDS) Brain Bank Criteria
* Demonstrate persistent motor fluctuations in spite of individually optimized treatment
* Subject must experience a minimum of 3 hours "Off" time

Exclusion Criteria:

* Subject's PD diagnosis is unclear or there is a suspicion that the subject has a Parkinsonian syndrome such as secondary Parkinsonism (e.g., caused by drugs, toxins, infectious agents, vascular disease, trauma, brain neoplasm), Parkinson-plus syndrome (e.g., Multiple System Atrophy, Progressive Supranuclear Palsy, Diffuse Lewy Body Disease, Corticobasilar Degeneration), or other neurodegenerative disease that might mimic the symptoms of PD.
* Subject has undergone neurosurgery for the treatment of Parkinson's disease
* Subject for whom the placement of a PEG-J tube for LCIG treatment is contraindicated or is considered a high risk for the PEG-J procedure according to the gastroenterology evaluation (e.g., pathological changes of the gastric wall, inability to bring the gastric wall and abdominal wall together, blood coagulation disorders, peritonitis, acute pancreatitis, paralytic ileus).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Benesh, BS, Study Director — AbbVie

REFERENCES:
- [Background] Standaert DG, Rodriguez RL, Slevin JT, Lobatz M, Eaton S, Chatamra K, Facheris MF, Hall C, Sail K, Jalundhwala YJ, Benesh J. Effect of Levodopa-carbidopa Intestinal Gel on Non-motor Symptoms in Patients with Advanced Parkinson's Disease. Mov Disord Clin Pract. 2017 Nov-Dec;4(6):829-837. doi: 10.1002/mdc3.12526. Epub 2017 Sep 20. PMID 29242809

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 12 sites in the United States that specialized in movement disorders. Participants were levodopa-responsive with advanced Parkinson's disease (PD) and persistent motor fluctuations despite attempts to optimize treatment with oral levodopa-carbidopa and other available anti-PD medications.
Pre-assignment Details: During screening participants converted their current daytime levodopa-carbidopa doses to oral levodopa-carbidopa 100/25 mg immediate release (LC-IR); other anti-PD medications could be continued, reduced or discontinued at the investigator's discretion. LC-IR and all other anti-PD treatments were discontinued at LCIG initiation.
Groups:
- Levodopa-Carbidopa Intestinal Gel (LCIG): Participants had a percutaneous endoscopic gastrostomy with jejunal extension (PEG-J) tube placement procedure performed on Day 1 and, at the discretion of the investigator, began initiation and titration of LCIG infusion. Dosing was determined individually. The starting total daily dose of LCIG was based solely on the daily dose of the oral levodopa taken immediately prior to Day 1 and was adjusted to obtain the optimal clinical response for the individual participant. Participants received treatment for up to 60 weeks; participants who completed their Week 60 visit before LCIG was commercially available had the option to extend their LCIG therapy, if in the opinion of the investigator, the participant would benefit from continued LCIG treatment.
Period: Overall Study
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Started | 39 (Enrolled participants who underwent the PEG-J placement procedure)
Received LCIG | 38
Completed | 28
Not Completed | 11
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 4
Not completed — Lack of Efficacy | 3
Not completed — Unable to Complete PEG Placement | 1

BASELINE CHARACTERISTICS:
Groups:
- Levodopa-Carbidopa Intestinal Gel: Participants had a PEG-J tube placement procedure performed on Day 1 and, at the discretion of the investigator, began initiation and titration of LCIG infusion. Dosing was determined individually and was adjusted to obtain the optimal clinical response for each participant. Participants received treatment for up to 60 weeks or until LCIG was commercially available.
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (10.23)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 17
  ≥ 65 years | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 36
  Black or African American | 1
  Asian | 2
  American Indian or Alaska Native | 0
  Native Hawaiian or other Pacific Islander | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 37
Duration of PD [Mean (Standard Deviation); unit: years] | 11.5 (5.34)
PD Symptoms Present [Count of Participants; unit: Participants]
  Bradykinesia | 37
  Muscular rigidity | 33
  Resting tremor | 25
  Postural instability | 22
Non-Motor Symptoms Scale (NMSS) Total Score [Mean (Standard Deviation); unit: units on a scale] — The NMSS assesses non-motor symptoms in Parkinson's Disease. It consists of 30 questions grouped into 9 domains: cardiovascular, sleep/fatigue, mood/cognition, perceptual problems/hallucinations, attention/memory, gastro-intestinal tract, urinary, sexual function, and miscellaneous. Severity is rated on a scale from 0 (none) to 3 (severe). Frequency is rated on a scale from 1 (rarely) to 4 (very frequent). The NMSS total score ranges from 0 to 360 with a lower score more desirable than a higher score. Baseline was the last measurement before the first dose of oral study drug. Population: Data are reported for the efficacy dataset which includes all participants who received at least 1 infusion of LCIG study drug and had a baseline and LCIG Treatment Period observation for at least one efficacy or health outcome measure.
  units on a scale
    number analyzed (Participants) | 38
    (all) | 48.3 (35.63)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in the Non-Motor Symptom Scale (NMSS) Total Score
Description: The NMSS measures the frequency and severity of a range of non-motor symptoms in Parkinson's Disease. It consists of 30 questions grouped into 9 domains: cardiovascular, sleep/fatigue, mood/cognition, perceptual problems/hallucinations, attention/memory, gastro-intestinal tract, urinary, sexual function, and miscellaneous (pain, taste/smell, weight change, excessive sweating). Severity is rated on a scale from 0 (none) to 3 (severe) and frequency is rated on a scale from 1 (rarely) to 4 (very frequent).
  Item scores are calculated as the product of severity and frequency; the total score is obtained by summing the item scores. The NMSS total score ranges from 0 to 360 with a lower score indicating fewer symptoms; a negative change from baseline indicates improvement in symptoms.
Time Frame: Baseline and Week 12
Population: The Efficacy dataset included all participants who received at least 1 infusion of LCIG study drug and had a baseline and LCIG Treatment Period observation for at least one efficacy or health outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 35
units on a scale | -17.6 (3.60)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel; The primary null hypothesis was no change in least-square (LS) mean, calculated using a mixed-effect repeated measures model (MMRM), for NMSS total score from baseline to Week 12. The statistical test was two-sided and the null hypothesis was rejected at the significance level of α = 0.050; Test type: Superiority or Other; p < 0.001, Mixed-effect Repeated Measures (MMRM); MMRM model included the fixed effects of study site and visit, with baseline score as a covariate, and the baseline-by-visit interaction

2. Secondary Outcome: Number of Participants Who Used Healthcare Resources During the First 4 Weeks
Description: Use of healthcare resources was assessed by the investigator using the Health Resource Utilization Questionnaire (HRUQ), a questionnaire developed by the Sponsor regarding the use of healthcare resources due to the participant's Parkinson's disease. The Week 4 version of the questionnaire addressed the following questions during the first four weeks after the PEG-J procedure:
  1. Has the subject had a visit to an emergency room?
  2. Has the subject had a visit to an urgent care?
  3. Has the subject had an outpatient visit to a neurologist?
  4. Has the subject had an outpatient visit to a gastroenterologist, surgeon, or interventional radiologist?
  5. Has the subject had an outpatient visit to a primary care physician?
  6. Has the subject called the nursing support line?
  7. Has the subject called a physician?
Time Frame: Weeks 1-4
Population: The Safety dataset included all participants who underwent the PEG-J placement procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
Participants
  Q1. Emergency Room Visit | 3
  Q2. Urgent Care Visit | 0
  Q3. Neurologist Visit | 6
  Q4. Gastroenterologist, Surgeon, Radiologist Visit | 11
  Q5. Primary Care Physician Visit | 8
  Q6. Called Nursing Support Line | 9
  Q7. Called Physician | 13

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events (AEs) related to treatment are those the investigator determined as having a reasonable possibility being related to study drug based on evidence to suggest a causal relationship between the study drug and the adverse event.
  A severe AE was defined as an adverse event that caused considerable interference with the participant's usual activities and might be incapacitating or life-threatening.
  Serious AEs were defined as those that were life-threatening or resulted in death, hospitalization or prolongation of hospitalization, a congenital anomaly, persistent or significant disability/incapacity, or important medical events requiring medical or surgical intervention to prevent a serious outcome.
Time Frame: Weeks 1-4 and Overall (from Week 1 through 30 days after the end of the LCIG Treatment Period; median duration of LCIG device exposure was 428 days)
Population: The Safety dataset
Measure: Count of Participants; unit: Participants
Groups:
- Week 1-4: Any adverse events that began or worsened in severity on or after the date of the first PEG-J placement procedure through week 4.
- Overall: Any adverse events that began or worsened in severity on or after the date of the first PEG-J placement procedure and no more than 30 days after the end of the LCIG Treatment Period.
Arm/Group | Week 1-4 | Overall
Number analyzed (Participants) | 39 | 39
Participants
  Any adverse event | 28 | 37
  AE related to LCIG | 26 | 35
  AE related to oral LC | 4 | 11
  Severe adverse event | 1 | 5
  Serious adverse event | 3 | 8
  AE leading to premature discontinuation | 1 | 5
  Gastrointestinal (GI) adverse event | 22 | 28
  Adverse event other than GI | 21 | 37
  Fatal adverse event | 0 | 1

4. Secondary Outcome: Number of Participants Who Used Healthcare Resources Through Week 60
Description: Use of healthcare resources was assessed by the investigator using the Health Resource Utilization Questionnaire (HRUQ), a questionnaire developed by the Sponsor regarding the use of healthcare resources due to the participant's Parkinson's disease. The standard version of the questionnaire addressed the following questions over the last 3 months:
  1. Has the subject had a visit to an emergency room?
  2. Has the subject had an outpatient visit to any of the following healthcare providers?
  3. Has the subject been visited in his or her place of residence by a health care professional?
  4. Has the subject received assistance from either of the following for their Parkinson's disease in their home?
  5. Has the subject needed to contact either of the following for immediate assistance related to their Parkinson's disease?
  6. Have family members or friends had to miss any paid work due to the subject's Parkinson's disease?
  7. Has the subject fallen during the past month?
Time Frame: Week 60
Population: Safety dataset with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 34
Participants
  Q1. Emergency Room Visit | 1
  Q2. Visit to Primary Care Physician | 18
  Q2. Visit to Gastroenterologist | 3
  Q2. Visit to Interventional Radiologist | 1
  Q2. Visit to Surgeon | 1
  Q2. Visit to Cardiologist | 1
  Q2. Visit to Endocrinologist | 0
  Q2. Visit to Immunologist | 0
  Q2. Visit to Internist | 1
  Q2. Visit to Psychiatrist | 0
  Q2. Visit to Urologist | 2
  Q2. Visit to Psychologist | 1
  Q2. Visit to Social Worker | 2
  Q2. Visit to Other Healthcare Provider | 10
  Q3. Visited by Physician | 0
  Q3. Visited by Nurse or Nurse Practitioner | 1
  Q3. Visited by Physical or Occupational Therapist | 0
  Q4. Received Unpaid Care From Family/Friend | 10
  Q4. Received Care From Paid Caregiver | 2
  Q5. Called 911 | 0
  Q5. Called Family/Friend | 1
  Q6. Family/Friends Missed Work | 2
  Q7. Fall During Past Month | 10

5. Secondary Outcome: Change From Baseline to Week 60 in the Non-Motor Symptom Scale (NMSS) Total Score
Description: as for outcome 1
Time Frame: Baseline and Week 60
Population: Efficacy dataset with available data at baseline and week 60
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 28
units on a scale | -11.8 (3.95)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel; Test type: Superiority or Other; p = 0.004, Mixed-effect Repeated Measures (MMRM); [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Change From Baseline in NMSS Cardiovascular Domain Score
Description: The NMSS measures the frequency and severity of a range of non-motor symptoms in Parkinson's Disease. It consists of 30 questions grouped into 9 domains: cardiovascular, sleep/fatigue, mood/cognition, perceptual problems/hallucinations, attention/memory, gastro-intestinal tract, urinary, sexual function, and miscellaneous (pain, taste/smell, weight change, excessive sweating). Severity is rated on a scale from 0 (none) to 3 (severe) and frequency is rated on a scale from 1 (rarely) to 4 (very frequent).
  Item scores are calculated as the product of severity and frequency; domain scores are obtained by summing the item scores. The NMSS cardiovascular including falls domain score ranges from 0 to 24 with a lower score indicating fewer symptoms; a negative change from baseline indicates improvement in symptoms.
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time points
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
units on a scale
  Week 12: number analyzed (Participants) | 35
  Week 12 | -0.2 (0.37)
  Week 60: number analyzed (Participants) | 28
  Week 60 | 0.5 (0.41)

7. Secondary Outcome: Change From Baseline in NMSS Sleep/Fatigue Domain Score
Description: The NMSS measures the frequency and severity of a range of non-motor symptoms in Parkinson's Disease. It consists of 30 questions grouped into 9 domains: cardiovascular, sleep/fatigue, mood/cognition, perceptual problems/hallucinations, attention/memory, gastro-intestinal tract, urinary, sexual function, and miscellaneous (pain, taste/smell, weight change, excessive sweating). Severity is rated on a scale from 0 (none) to 3 (severe) and frequency is rated on a scale from 1 (rarely) to 4 (very frequent).
  Item scores are calculated as the product of severity and frequency; domain scores are obtained by summing the item scores. The NMSS sleep/fatigue domain score ranges from 0 to 48 with a lower score indicating fewer symptoms; a negative change from baseline indicates improvement in symptoms.
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
units on a scale
  Week 12: number analyzed (Participants) | 35
  Week 12 | -6.0 (1.17)
  Week 60: number analyzed (Participants) | 28
  Week 60 | -5.4 (1.29)

8. Secondary Outcome: Change From Baseline in NMSS Mood/Cognition Domain Score
Description: The NMSS measures the frequency and severity of a range of non-motor symptoms in Parkinson's Disease. It consists of 30 questions grouped into 9 domains: cardiovascular, sleep/fatigue, mood/cognition, perceptual problems/hallucinations, attention/memory, gastro-intestinal tract, urinary, sexual function, and miscellaneous (pain, taste/smell, weight change, excessive sweating). Severity is rated on a scale from 0 (none) to 3 (severe) and frequency is rated on a scale from 1 (rarely) to 4 (very frequent).
  Item scores are calculated as the product of severity and frequency; domain scores are obtained by summing the item scores. The NMSS mood/cognition domain score ranges from 0 to 72 with a lower score indicating fewer symptoms; a negative change from baseline indicates improvement in symptoms.
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
units on a scale
  Week 12: number analyzed (Participants) | 35
  Week 12 | 0.0 (1.12)
  Week 60: number analyzed (Participants) | 28
  Week 60 | 0.5 (1.24)

9. Secondary Outcome: Change From Baseline in NMSS Perceptual Problems/Hallucinations Domain Score
Description: The NMSS measures the frequency and severity of a range of non-motor symptoms in Parkinson's Disease. It consists of 30 questions grouped into 9 domains: cardiovascular, sleep/fatigue, mood/cognition, perceptual problems/hallucinations, attention/memory, gastro-intestinal tract, urinary, sexual function, and miscellaneous (pain, taste/smell, weight change, excessive sweating). Severity is rated on a scale from 0 (none) to 3 (severe) and frequency is rated on a scale from 1 (rarely) to 4 (very frequent).
  Item scores are calculated as the product of severity and frequency; domain scores are obtained by summing the item scores. The NMSS perceptual problems/hallucinations domain score ranges from 0 to 36 with a lower score indicating fewer symptoms; a negative change from baseline indicates improvement in symptoms.
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
units on a scale
  Week 12: number analyzed (Participants) | 35
  Week 12 | -0.5 (0.38)
  Week 60: number analyzed (Participants) | 28
  Week 60 | 0.4 (0.43)

10. Secondary Outcome: Change From Baseline in NMSS Attention/Memory Domain Score
Description: The NMSS measures the frequency and severity of a range of non-motor symptoms in Parkinson's Disease. It consists of 30 questions grouped into 9 domains: cardiovascular, sleep/fatigue, mood/cognition, perceptual problems/hallucinations, attention/memory, gastro-intestinal tract, urinary, sexual function, and miscellaneous (pain, taste/smell, weight change, excessive sweating). Severity is rated on a scale from 0 (none) to 3 (severe) and frequency is rated on a scale from 1 (rarely) to 4 (very frequent).
  Item scores are calculated as the product of severity and frequency; domain scores are obtained by summing the item scores. The NMSS attention/memory domain score ranges from 0 to 36 with a lower score indicating fewer symptoms; a negative change from baseline indicates improvement in symptoms.
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
units on a scale
  Week 12: number analyzed (Participants) | 35
  Week 12 | -2.1 (0.80)
  Week 60: number analyzed (Participants) | 28
  Week 60 | -2.2 (0.87)

11. Secondary Outcome: Change From Baseline in NMSS Gastrointestinal Tract Domain Score
Description: The NMSS measures the frequency and severity of a range of non-motor symptoms in Parkinson's Disease. It consists of 30 questions grouped into 9 domains: cardiovascular, sleep/fatigue, mood/cognition, perceptual problems/hallucinations, attention/memory, gastro-intestinal tract, urinary, sexual function, and miscellaneous (pain, taste/smell, weight change, excessive sweating). Severity is rated on a scale from 0 (none) to 3 (severe) and frequency is rated on a scale from 1 (rarely) to 4 (very frequent).
  Item scores are calculated as the product of severity and frequency; domain scores are obtained by summing the item scores. The NMSS gastrointestinal tract domain score ranges from 0 to 36 with a lower score indicating fewer symptoms; a negative change from baseline indicates improvement in symptoms.
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
units on a scale
  Week 12: number analyzed (Participants) | 35
  Week 12 | -2.0 (0.60)
  Week 60: number analyzed (Participants) | 28
  Week 60 | -1.9 (0.67)

12. Secondary Outcome: Change From Baseline in NMSS Urinary Domain Score
Description: The NMSS measures the frequency and severity of a range of non-motor symptoms in Parkinson's Disease. It consists of 30 questions grouped into 9 domains: cardiovascular, sleep/fatigue, mood/cognition, perceptual problems/hallucinations, attention/memory, gastro-intestinal tract, urinary, sexual function, and miscellaneous (pain, taste/smell, weight change, excessive sweating). Severity is rated on a scale from 0 (none) to 3 (severe) and frequency is rated on a scale from 1 (rarely) to 4 (very frequent).
  Item scores are calculated as the product of severity and frequency; domain scores are obtained by summing the item scores. The NMSS urinary domain score ranges from 0 to 36 with a lower score indicating fewer symptoms; a negative change from baseline indicates improvement in symptoms.
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
units on a scale
  Week 12: number analyzed (Participants) | 35
  Week 12 | -2.2 (1.07)
  Week 60: number analyzed (Participants) | 28
  Week 60 | 0.1 (1.19)

13. Secondary Outcome: Change From Baseline in NMSS Sexual Function Domain Score
Description: The NMSS measures the frequency and severity of a range of non-motor symptoms in Parkinson's Disease. It consists of 30 questions grouped into 9 domains: cardiovascular, sleep/fatigue, mood/cognition, perceptual problems/hallucinations, attention/memory, gastro-intestinal tract, urinary, sexual function, and miscellaneous (pain, taste/smell, weight change, excessive sweating). Severity is rated on a scale from 0 (none) to 3 (severe) and frequency is rated on a scale from 1 (rarely) to 4 (very frequent).
  Item scores are calculated as the product of severity and frequency; domain scores are obtained by summing the item scores. The NMSS sexual function domain score ranges from 0 to 24 with a lower score indicating fewer symptoms; a negative change from baseline indicates improvement in symptoms.
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
units on a scale
  Week 12: number analyzed (Participants) | 35
  Week 12 | -1.8 (0.42)
  Week 60: number analyzed (Participants) | 28
  Week 60 | -1.1 (0.47)

14. Secondary Outcome: Change From Baseline in NMSS Miscellaneous Domain Score
Description: The NMSS measures the frequency and severity of a range of non-motor symptoms in Parkinson's Disease. It consists of 30 questions grouped into 9 domains: cardiovascular, sleep/fatigue, mood/cognition, perceptual problems/hallucinations, attention/memory, gastro-intestinal tract, urinary, sexual function, and miscellaneous (pain, taste/smell, weight change, excessive sweating). Severity is rated on a scale from 0 (none) to 3 (severe) and frequency is rated on a scale from 1 (rarely) to 4 (very frequent).
  Item scores are calculated as the product of severity and frequency; domain scores are obtained by summing the item scores. The NMSS miscellaneous domain score ranges from 0 to 48 with a lower score indicating fewer symptoms; a negative change from baseline indicates improvement in symptoms.
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
units on a scale
  Week 12: number analyzed (Participants) | 35
  Week 12 | -3.4 (1.00)
  Week 60: number analyzed (Participants) | 28
  Week 60 | -3.4 (1.11)

15. Secondary Outcome: Change From Baseline in Mean Daily Normalized "Off" Time Based on Parkinson's Disease Diary
Description: The Parkinson's Disease Diary was completed by the participant for 3 consecutive days prior to each visit for the full 24 hours of each day. Participants recorded whether they had been "On," "Off," or "Asleep" and the severity of their dyskinesias (troublesome or not troublesome) for each 30-minute period during their normal waking time and upon awakening from time asleep.
  "Off" time was defined as time when medication has worn off and was no longer providing benefit with regard to mobility, slowness, and stiffness.
  Parkinson's Disease Diary times were normalized to a 16-hour waking time to account for variation in participants' sleep time. Normalized PD Diary times at a given visit were calculated as the average normalized time from the PD Diary for the 3 days prior to the visit.
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
hours
  Week 12: number analyzed (Participants) | 32
  Week 12 | -4.1 (0.39)
  Week 60: number analyzed (Participants) | 21
  Week 60 | -4.9 (0.48)

16. Secondary Outcome: Change From Baseline in Mean Daily Normalized "On" Time Without Troublesome Dyskinesia Based on PD Diary
Description: The PD Diary was completed by the participant for 3 consecutive days prior to each visit. Participants recorded whether they had been "On," "Off," or "Asleep" and the severity of their dyskinesias (troublesome or not troublesome) for each 30-minute period during their normal waking time and upon awakening from sleep.
  "On" was defined as time when medication was providing benefit with regard to mobility, slowness, and stiffness. "On" time without troublesome dyskinesia is a composite of "On" time without dyskinesia (involuntary twisting, turning movements which are an effect of medication) plus "On" time with non-troublesome dyskinesia (dyskinesia that does not interfere with function or cause meaningful discomfort).
  PD Diary times were normalized to a 16-hour waking time to account for variation in participants' sleep time. Normalized PD Diary times at a given visit were calculated as the average normalized time from the PD Diary for the 3 days prior to the visit.
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
hours
  Week 12: number analyzed (Participants) | 32
  Week 12 | 3.7 (0.48)
  Week 60: number analyzed (Participants) | 21
  Week 60 | 4.3 (0.58)

17. Secondary Outcome: Change From Baseline for Unified Parkinson's Disease Rating Scale (UPDRS) Total Score
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) is an investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The UPDRS assessment was performed by an approved, trained rater.
  The UPDRS was made up of the following sections:
  * Part I - Mentation, Behavior, and Mood
  * Part II - Activities of Daily Living
  * Part III - Motor Examination
  * Part IV - Complications of Therapy (including dyskinesias)
  * Part V - Modified Hoehn and Yahr Staging
  The Total UPDRS score includes 31 items contributing to three subscales: (I) Mentation, Behavior, and Mood; (II) Activities of Daily Living; and (III) Motor Examination. Each question is answered on a scale from 0 (None) to 4 (Severe); Some questions require multiple grades assigned to each extremity. The UPDRS Total score was computed as the sum of these 3 UPDRS subscales and ranged from 0 to 176, with 176 representing the worst (total) disability, and 0 no disability.
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at baseline (37) and each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 37
units on a scale
  Week 12: number analyzed (Participants) | 34
  Week 12 | -11.4 (1.67)
  Week 60: number analyzed (Participants) | 28
  Week 60 | -7.7 (2.26)

18. Secondary Outcome: Change From Baseline in UPDRS Part I: Mentation, Behavior, and Mood Score
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) is an investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The UPDRS assessment was performed by an approved, trained rater.
  The UPDRS was made up of the following sections:
  * Part I - Mentation, Behavior, and Mood
  * Part II - Activities of Daily Living
  * Part III - Motor Examination
  * Part IV - Complications of Therapy (including dyskinesias)
  * Part V - Modified Hoehn and Yahr Staging
  The mentation, behavior, and mood score includes 4 items addressing intellectual impairment, thought disorder, motivation/initiative, and depression. Each question is answered on a scale from 0 (None) to 4 (Severe). The UPDRS Part I: mentation, behavior, and mood score was computed as the sum of these items and ranged from 0 (not affected) to 16 (most severely affected).
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at baseline (37) and each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 37
units on a scale
  Week 12: number analyzed (Participants) | 34
  Week 12 | -0.3 (0.31)
  Week 60: number analyzed (Participants) | 28
  Week 60 | -0.1 (0.26)

19. Secondary Outcome: Change From Baseline in UPDRS Part II: Activities of Daily Living (ADL) Score
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) is an investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The UPDRS assessment was performed by an approved, trained rater.
  The UPDRS was made up of the following sections:
  * Part I - Mentation, Behavior, and Mood
  * Part II - Activities of Daily Living
  * Part III - Motor Examination
  * Part IV - Complications of Therapy (including dyskinesias)
  * Part V - Modified Hoehn and Yahr Staging
  The activities of daily living score includes 13 items addressing speech, salivation, swallowing, handwriting, cutting food, dressing, hygiene, turning in bed, falling, freezing, walking, tremor, and sensory complaints. Each question is answered on a scale from 0 (Normal) to 4 (Severe). The UPDRS Part II: activities of daily living score was computed as the sum of these items and ranged from 0 (not affected) to 52 (most severely affected).
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at baseline (37) and at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 37
units on a scale
  Week 12: number analyzed (Participants) | 34
  Week 12 | -5.5 (0.89)
  Week 60: number analyzed (Participants) | 28
  Week 60 | -4.7 (0.92)

20. Secondary Outcome: Change From Baseline in UPDRS Part III: Motor Examination Score
Description: The UPDRS is an investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The UPDRS assessment was performed by an approved, trained rater.
  The UPDRS was made up of the following sections:
  * Part I - Mentation, Behavior, and Mood
  * Part II - Activities of Daily Living
  * Part III - Motor Examination
  * Part IV - Complications of Therapy (including dyskinesias)
  * Part V - Modified Hoehn and Yahr Staging
  The motor examination score includes 17 items addressing speech, facial expression, tremor at rest, action tremor, rigidity, finger taps, hand movements, hand pronation and supination, leg agility, arising from chair, posture, gait, postural stability, and body bradykinesia. Each question is answered on a scale from 0 (Normal) to 4 (Severe), some items include multiple grades for each extremity. The UPDRS Part III: motor examination score was computed as the sum of these items and ranged from 0 (not affected) to 108 (most severely affected).
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at baseline (37) and at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 37
units on a scale
  Week 12: number analyzed (Participants) | 34
  Week 12 | -5.6 (1.19)
  Week 60: number analyzed (Participants) | 28
  Week 60 | -3.6 (1.49)

21. Secondary Outcome: Change From Baseline in UPDRS Part IV: Complications of Therapy Score
Description: The UPDRS is an investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The UPDRS assessment was performed by an approved, trained rater.
  The UPDRS was made up of the following sections:
  * Part I - Mentation, Behavior, and Mood
  * Part II - Activities of Daily Living
  * Part III - Motor Examination
  * Part IV - Complications of Therapy (including dyskinesias)
  * Part V - Modified Hoehn and Yahr Staging
  The complications of therapy section includes 11 items addressing dyskinesia duration, disability, and pain, early morning dystonia, "offs"-predictable, "offs"-unpredictable, "offs"-sudden, "offs"-duration, anorexia-nausea-vomiting, sleep disturbance, and symptomatic orthostasis. Four questions are answered on a scale from 0 (Normal) to 4 (Severe) and seven on a binary scale where 0=No and 1=Yes. The UPDRS Part IV: complications of therapy score was computed as the sum of these items and ranged from 0 (not affected) to 23 (most severely affected).
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
units on a scale
  Week 12: number analyzed (Participants) | 35
  Week 12 | -3.5 (0.44)
  Week 60: number analyzed (Participants) | 28
  Week 60 | -2.9 (0.57)

22. Secondary Outcome: Change From Baseline in UPDRS Dyskinesia Items Score
Description: The UPDRS is an investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The UPDRS assessment was performed by an approved, trained rater.
  The UPDRS was made up of the following sections:
  * Part I - Mentation, Behavior, and Mood
  * Part II - Activities of Daily Living
  * Part III - Motor Examination
  * Part IV - Complications of Therapy (including dyskinesias)
  * Part V - Modified Hoehn and Yahr Staging
  The dyskinesia items score includes questions 32, 33 and 34 from the complications of therapy section of the UPDRS which address dyskinesia duration, disability, and pain. Each question was answered on a scale from 0 (Normal) to 4 (Severe); the UPDRS dyskinesia items score was computed as the sum of these items and ranged from 0 (not affected) to 12 (most severely affected).
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
units on a scale
  Week 12: number analyzed (Participants) | 35
  Week 12 | -1.1 (0.28)
  Week 60: number analyzed (Participants) | 28
  Week 60 | -0.6 (0.36)

23. Secondary Outcome: Change From Baseline in UPDRS Part V: Modified Hoehn and Yahr Staging Score
Description: The UPDRS is an investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The UPDRS assessment was performed by an approved, trained rater.
  The UPDRS was made up of the following sections:
  * Part I - Mentation, Behavior, and Mood
  * Part II - Activities of Daily Living
  * Part III - Motor Examination
  * Part IV - Complications of Therapy (including dyskinesias)
  * Part V - Modified Hoehn and Yahr Staging
  The modified Hoehn and Yahr scale is as follows:
  * Stage 0: No signs of disease
  * Stage 1.0: Symptoms are very mild; unilateral involvement only
  * Stage 1.5: Unilateral and axial involvement
  * Stage 2: Bilateral involvement without impairment of balance
  * Stage 2.5: Mild bilateral disease with recovery on pull test
  * Stage 3: Mild to moderate bilateral disease; some postural instability; physically independent
  * Stage 4: Severe disability; still able to walk or stand unassisted
  * Stage 5: Wheelchair bound or bedridden unless aided
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
units on a scale
  Week 12: number analyzed (Participants) | 35
  Week 12 | -0.2 (0.10)
  Week 60: number analyzed (Participants) | 28
  Week 60 | -0.2 (0.12)

24. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire-39 Item (PDQ-39) Summary Index
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing eight domains of health (mobility [10 items], activities of daily living [six items], emotional wellbeing [six items], stigma [four items], communication [three items] and bodily discomfort [three items]) which subjects consider to be adversely affected by the disease. Each item is scored on the following 5-point scale: 0 = Never, 1 = Occasionally, 2 = Sometimes, 3 = Often, 4 = Always (or cannot do at all, if applicable).
  The PDQ-39 Summary Index (PDQ-SI) is the sum of all answers divided by the highest score possible (i.e., number of answers multiplied by 4) which is multiplied by 100 to put the score on a 0 - 100 scale where lower scores indicate a better perceived health status and higher scores are associated with the more severe symptoms of the disease such as tremors and stiffness.
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
units on a scale
  Week 12: number analyzed (Participants) | 34
  Week 12 | -11.2 (2.75)
  Week 60: number analyzed (Participants) | 28
  Week 60 | -10.2 (2.63)

25. Secondary Outcome: Change From Baseline in PDQ-39 Mobility Domain Score
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing eight domains of health (mobility [10 items], activities of daily living [six items], emotional wellbeing [six items], stigma [four items], communication [three items] and bodily discomfort [three items]) which subjects consider to be adversely affected by the disease. Each item is scored on the following 5-point scale: 0 = Never, 1 = Occasionally, 2 = Sometimes, 3 = Often, 4 = Always (or cannot do at all, if applicable).
  Domain scores are calculated by summing the answers to the questions in the domain, dividing by the highest score possible and then multiplying by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status and higher scores are associated with the more severe symptoms of the disease such as tremors and stiffness.
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
units on a scale
  Week 12: number analyzed (Participants) | 34
  Week 12 | -18.5 (4.39)
  Week 60: number analyzed (Participants) | 28
  Week 60 | -19.4 (4.21)

26. Secondary Outcome: Change From Baseline in PDQ-39 Activities of Daily Living Domain Score
Description: as for outcome 25
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
units on a scale
  Week 12: number analyzed (Participants) | 34
  Week 12 | -12.1 (4.43)
  Week 60: number analyzed (Participants) | 28
  Week 60 | -11.9 (4.23)

27. Secondary Outcome: Change From Baseline in PDQ-39 Emotional Well-Being Domain Score
Description: as for outcome 25
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
units on a scale
  Week 12: number analyzed (Participants) | 34
  Week 12 | -4.9 (3.14)
  Week 60: number analyzed (Participants) | 26
  Week 60 | -6.6 (3.74)

28. Secondary Outcome: Change From Baseline in PDQ-39 Stigma Domain Score
Description: as for outcome 25
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
units on a scale
  Week 12: number analyzed (Participants) | 34
  Week 12 | -9.5 (2.38)
  Week 60: number analyzed (Participants) | 28
  Week 60 | -5.4 (3.01)

29. Secondary Outcome: Change From Baseline in PDQ-39 Social Support Domain Score
Description: as for outcome 25
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
units on a scale
  Week 12: number analyzed (Participants) | 34
  Week 12 | 1.6 (2.62)
  Week 60: number analyzed (Participants) | 28
  Week 60 | 3.3 (2.95)

30. Secondary Outcome: Change From Baseline in PDQ-39 Cognition Domain Score
Description: as for outcome 25
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
units on a scale
  Week 12: number analyzed (Participants) | 34
  Week 12 | -8.4 (2.23)
  Week 60: number analyzed (Participants) | 28
  Week 60 | -7.3 (2.00)

31. Secondary Outcome: Change From Baseline in PDQ-39 Communication Domain Score
Description: as for outcome 25
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
units on a scale
  Week 12: number analyzed (Participants) | 34
  Week 12 | -13.0 (3.24)
  Week 60: number analyzed (Participants) | 27
  Week 60 | -10.8 (2.59)

32. Secondary Outcome: Change From Baseline in PDQ-39 Bodily Discomfort Domain Score
Description: as for outcome 25
Time Frame: Baseline and Week 12 and Week 60
Population: Efficacy dataset with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
units on a scale
  Week 12: number analyzed (Participants) | 33
  Week 12 | -9.6 (4.40)
  Week 60: number analyzed (Participants) | 28
  Week 60 | -3.8 (3.65)

33. Secondary Outcome: Percentage of Participants With a Patient Global Impression of Change (PGIC) Response of Improved
Description: The PGIC is a 7-point response scale. Participants were asked to rate their change in status using the following 7-point scale:
  1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse.
  The responses of "Very much improved," "Much improved" and "Minimally improved" on the PGIC were used to define responders.
Time Frame: Week 12 and Week 60
Population: Efficacy dataset
Measure: Number; unit: percentage of participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 38
percentage of participants
  Week 12 | 78.9
  Week 60 | 71.1

34. Secondary Outcome: Treatment Satisfaction Questionnaire Scores
Description: The Treatment Satisfaction Questionnaire (TSQ) is a single item instrument developed by the Sponsor on which the participant indicated their level of satisfaction or dissatisfaction with their PD treatment. The responses are recorded on a Likert-type scale (Very Satisfied, Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Dissatisfied, Very Dissatisfied).
Time Frame: Week 12 and Week 60
Population: Efficacy dataset
Measure: Count of Participants; unit: Participants
Arm/Group | Week 12 | Week 60
Number analyzed (Participants) | 38 | 38
Participants
  Very satisfied | 15 | 14
  Satisfied | 14 | 9
  Somewhat satisfied | 4 | 3
  Somewhat dissatisfied | 1 | 1
  Dissatisfied | 1 | 0
  Very dissatisfied | 0 | 1
  Missing | 3 | 10

35. Secondary Outcome: Change From Baseline in Health-related Productivity
Description: The Health-Related Productivity Questionnaire (HRPQ) is a generic measure of the impact of disease on the ability of the participant to be productive at paid employment or at performance of household chores. Questions inquire about the amount of time they were scheduled/planned to work, the number of the scheduled/planned hours they were able to work and their ability to be productive for the hours of work they did perform.
  Absenteeism: Number of hours not worked due to PD or it's treatments;
  Presenteeism: Number of hours of lost productivity while at work due to PD or it's treatments;
  Total hours lost: Number of hours lost due to absenteeism and presenteeism
Time Frame: Baseline, Week 12 and Week 60
Population: Efficacy dataset with available data. Workplace hours lost is calculated for participants who were employed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Week 12 | Week 60
Number analyzed (Participants) | 28 | 28
hours
  Workplace Work Lost - Absenteeism: number analyzed (Participants) | 7 | 6
  Workplace Work Lost - Absenteeism | -2.1 (4.63) | -5.2 (6.27)
  Household Work Lost - Absenteeism: number analyzed (Participants) | 23 | 21
  Household Work Lost - Absenteeism | -3.5 (11.19) | -1.9 (8.38)
  Workplace Work Lost - Presenteeism: number analyzed (Participants) | 7 | 6
  Workplace Work Lost - Presenteeism | -0.8 (13.04) | -0.3 (3.87)
  Household Work Lost - Presenteeism: number analyzed (Participants) | 23 | 21
  Household Work Lost - Presenteeism | -1.8 (6.42) | -1.9 (5.42)
  Total Workplace Work Lost: number analyzed (Participants) | 7 | 6
  Total Workplace Work Lost | -3.0 (8.87) | -5.5 (4.50)
  Total Household Work Lost: number analyzed (Participants) | 23 | 21
  Total Household Work Lost | -5.3 (15.69) | -3.8 (11.26)

36. Secondary Outcome: Change From Baseline in Cambridge Neuropsychological Test Automated Battery (CANTAB) Spatial Working Memory Between Errors Score at Week 12
Description: CANTAB is a computer-based test of the participant's ability to retain spatial information and to manipulate remembered items in working memory. The Spatial Working Memory module requires that subjects find a blue token in a series of displayed boxes and use these to fill up an empty column, while not returning to boxes where a blue token has been previously found. The between errors score is the number of times the participant revisited a box in which a token was previously found; errors are calculated for 4-, 6-, and 8-box trials. Higher numbers indicate poorer performance.
Time Frame: Baseline and Week 12
Population: Efficacy dataset with available data
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 18
errors | -0.6 (7.73)

37. Secondary Outcome: Change From Baseline in CANTAB Spatial Working Memory Strategy Score at Week 12
Description: CANTAB is a computer-based test of the participant's ability to retain spatial information and to manipulate remembered items in working memory. The Spatial Working Memory module requires that subjects find a blue token in a series of displayed boxes and use these to fill up an empty column, while not returning to boxes where a blue token has been previously found. The Strategy score represents the number of times a participant begins a search with the same box for 6- and 8-box problems. Minimum score is 8 and maximum score is 56. Higher numbers indicate poorer performance.
Time Frame: Baseline and Week 12
Population: Efficacy dataset with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 18
units on a scale | 0.8 (2.31)

38. Secondary Outcome: Change From Baseline in Controlled Oral Word Association Test (COWAT) Verbal Fluency Scores at Week 60
Description: Letter fluency was assessed using a paper and pen test, in which participants were asked to generate as many words as possible in 60 seconds, starting with the letters F, A, or S.
  The COWAT All Letters score is the number of words recalled in all post-baseline assessments, regardless of letter used.
  The COWAT Baseline Letter score is the number of words recalled in post-baseline assessments that used the same letter as at Baseline.
Time Frame: Baseline and Week 60
Population: Efficacy dataset with available data
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Number analyzed (Participants) | 31
words
  All Letters Score: number analyzed (Participants) | 20
  All Letters Score | -0.5 (4.80)
  Baseline Letter Score: number analyzed (Participants) | 12
  Baseline Letter Score | -1.8 (4.03)

ADVERSE EVENTS:
Time Frame: Weeks 1-4 and Overall (from Week 1 through 30 days after the end of the LCIG Treatment Period; median duration of LCIG device exposure was 428 days).
Arm/Group | Levodopa-Carbidopa Intestinal Gel
Serious Adverse Events (participants affected / at risk) | 8/39
Other Adverse Events (participants affected / at risk) | 36/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levodopa-Carbidopa Intestinal Gel (N=39)
ATRIAL FIBRILLATION (Cardiac disorders) | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1
INTERNAL HERNIA (Gastrointestinal disorders) | 1
PERITONITIS (Infections and infestations) | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
RADICULOPATHY (Nervous system disorders) | 1
SEDATION (Nervous system disorders) | 1
ANXIETY (Psychiatric disorders) | 1
MAJOR DEPRESSION (Psychiatric disorders) | 1
SUICIDAL IDEATION (Psychiatric disorders) | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levodopa-Carbidopa Intestinal Gel (N=39)
ANAEMIA (Blood and lymphatic system disorders) | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1
TACHYCARDIA (Cardiac disorders) | 1
EAR PAIN (Ear and labyrinth disorders) | 1
AMAUROSIS FUGAX (Eye disorders) | 1
CATARACT (Eye disorders) | 1
DRY EYE (Eye disorders) | 1
MACULAR DEGENERATION (Eye disorders) | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 3
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1
ABDOMINAL TENDERNESS (Gastrointestinal disorders) | 1
BARRETT'S OESOPHAGUS (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 3
DENTAL CARIES (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 2
DIVERTICULUM (Gastrointestinal disorders) | 1
DRY MOUTH (Gastrointestinal disorders) | 2
DYSPHAGIA (Gastrointestinal disorders) | 1
FAECES SOFT (Gastrointestinal disorders) | 1
FLATULENCE (Gastrointestinal disorders) | 4
GASTRIC POLYPS (Gastrointestinal disorders) | 1
GASTRITIS (Gastrointestinal disorders) | 1
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2
HIATUS HERNIA (Gastrointestinal disorders) | 1
ILEUS (Gastrointestinal disorders) | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 2
NAUSEA (Gastrointestinal disorders) | 4
PANCREATIC MASS (Gastrointestinal disorders) | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1
TOOTHACHE (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 1
ADMINISTRATION SITE ODOUR (General disorders) | 1
APPLICATION SITE IRRITATION (General disorders) | 1
CATHETER SITE DERMATITIS (General disorders) | 1
CATHETER SITE ERYTHEMA (General disorders) | 1
CATHETER SITE HAEMATOMA (General disorders) | 1
CATHETER SITE PAIN (General disorders) | 1
CYST (General disorders) | 1
DEVICE DISLOCATION (General disorders) | 2
DRUG EFFECT DECREASED (General disorders) | 1
FATIGUE (General disorders) | 1
FEELING COLD (General disorders) | 1
INFLAMMATION (General disorders) | 1
NON-CARDIAC CHEST PAIN (General disorders) | 1
OEDEMA PERIPHERAL (General disorders) | 1
PAIN (General disorders) | 2
PYREXIA (General disorders) | 1
BILE DUCT STONE (Hepatobiliary disorders) | 1
BRONCHITIS (Infections and infestations) | 1
CYSTITIS (Infections and infestations) | 1
LOCALISED INFECTION (Infections and infestations) | 2
PNEUMONIA (Infections and infestations) | 2
PYODERMA (Infections and infestations) | 1
STOMA SITE ABSCESS (Infections and infestations) | 2
STOMA SITE INFECTION (Infections and infestations) | 11
TOOTH INFECTION (Infections and infestations) | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 6
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 1
AGITATION POSTOPERATIVE (Injury, poisoning and procedural complications) | 1
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 1
FALL (Injury, poisoning and procedural complications) | 7
LACERATION (Injury, poisoning and procedural complications) | 3
OESOPHAGEAL INJURY (Injury, poisoning and procedural complications) | 1
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 13
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1
SKIN ABRASION (Injury, poisoning and procedural complications) | 2
STERNAL FRACTURE (Injury, poisoning and procedural complications) | 1
STOMA SITE DISCHARGE (Injury, poisoning and procedural complications) | 3
STOMA SITE ERYTHEMA (Injury, poisoning and procedural complications) | 8
STOMA SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 3
STOMA SITE INFLAMMATION (Injury, poisoning and procedural complications) | 1
STOMA SITE IRRITATION (Injury, poisoning and procedural complications) | 4
STOMA SITE PAIN (Injury, poisoning and procedural complications) | 9
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1
ULNAR NERVE INJURY (Injury, poisoning and procedural complications) | 1
BLOOD CHOLESTEROL INCREASED (Investigations) | 1
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1
VIBRATION TEST ABNORMAL (Investigations) | 1
VITAMIN B12 DECREASED (Investigations) | 2
VITAMIN B6 DECREASED (Investigations) | 2
VITAMIN B6 INCREASED (Investigations) | 1
WEIGHT DECREASED (Investigations) | 7
DECREASED APPETITE (Metabolism and nutrition disorders) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 2
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 1
VITAMIN B12 DEFICIENCY (Metabolism and nutrition disorders) | 3
VITAMIN B6 DEFICIENCY (Metabolism and nutrition disorders) | 4
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2
BURSITIS (Musculoskeletal and connective tissue disorders) | 1
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1
LIMB DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 2
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
HAEMANGIOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
AKINESIA (Nervous system disorders) | 1
AREFLEXIA (Nervous system disorders) | 1
BALANCE DISORDER (Nervous system disorders) | 1
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 1
COGNITIVE DISORDER (Nervous system disorders) | 3
DEMENTIA (Nervous system disorders) | 1
DIZZINESS (Nervous system disorders) | 1
DROOLING (Nervous system disorders) | 1
DYSGEUSIA (Nervous system disorders) | 1
DYSKINESIA (Nervous system disorders) | 3
DYSTONIA (Nervous system disorders) | 1
ENCEPHALOPATHY (Nervous system disorders) | 1
HYPOAESTHESIA (Nervous system disorders) | 2
LOSS OF PROPRIOCEPTION (Nervous system disorders) | 1
LUMBAR RADICULOPATHY (Nervous system disorders) | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1
PARAESTHESIA (Nervous system disorders) | 1
PARKINSON'S DISEASE (Nervous system disorders) | 3
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2
PRESYNCOPE (Nervous system disorders) | 1
RESTLESS LEGS SYNDROME (Nervous system disorders) | 1
SOMNOLENCE (Nervous system disorders) | 1
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 1
ANXIETY (Psychiatric disorders) | 7
APATHY (Psychiatric disorders) | 1
DELUSION (Psychiatric disorders) | 1
DEPRESSED MOOD (Psychiatric disorders) | 1
DEPRESSION (Psychiatric disorders) | 3
HALLUCINATION (Psychiatric disorders) | 3
HYPOMANIA (Psychiatric disorders) | 1
INSOMNIA (Psychiatric disorders) | 3
SLEEP DISORDER (Psychiatric disorders) | 1
BLADDER OUTLET OBSTRUCTION (Renal and urinary disorders) | 1
BLADDER SPASM (Renal and urinary disorders) | 1
DYSURIA (Renal and urinary disorders) | 1
MICTURITION URGENCY (Renal and urinary disorders) | 1
NOCTURIA (Renal and urinary disorders) | 1
POLLAKIURIA (Renal and urinary disorders) | 1
RENAL CYST (Renal and urinary disorders) | 1
RENAL FAILURE (Renal and urinary disorders) | 1
URETHRAL HAEMORRHAGE (Renal and urinary disorders) | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 1
URINARY RETENTION (Renal and urinary disorders) | 1
PROSTATOMEGALY (Reproductive system and breast disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 1
YAWNING (Respiratory, thoracic and mediastinal disorders) | 1
BLISTER (Skin and subcutaneous tissue disorders) | 1
COLD SWEAT (Skin and subcutaneous tissue disorders) | 1
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 1
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 1
EXCESSIVE GRANULATION TISSUE (Skin and subcutaneous tissue disorders) | 4
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 2
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 1
LENTIGO (Skin and subcutaneous tissue disorders) | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 1
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1
SKIN LESION (Skin and subcutaneous tissue disorders) | 2
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.